CLINICAL TRIAL: NCT04994379
Title: Investigating the Effect of the Intensity of Primary Motor Cortex Cathodal TDCS on Appetite; a Double-blind Sham-controlled Study
Brief Title: Investigating the Effects of Intensity of Transcranial Direct Current Stimulation on Subjective Appetite
Acronym: tDCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Working conditions.
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Abed Hadipour Lakmehsari, Principal Investigator, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Tongue Motor Cortex
Record Dates: First submitted 2021-07-01; First posted 2021-08-06 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: Perceived appetite; tDCS; Submental muscle; M1

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of the three groups of active 1 mA, active 1.5 mA, or the sham group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1 mA tDCS (Experimental): Participants receive the stimulation with an intensity of 1 mA.
  Interventions: Device: 1 mA tDCS
- 1.5 mA tDCS (Experimental): Participants receive the stimulation with an intensity of 1.5 mA.
  Interventions: Device: 1.5 mA tDCS
- Sham tDCS (Sham Comparator): Participants receive the sham stimulation (zero electric current after a short initial increase).
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: 1 mA tDCS — One session with stimulation intensity of 1 mA.
  Arms: 1 mA tDCS
Device: 1.5 mA tDCS — One session with stimulation intensity of 1.5 mA.
  Arms: 1.5 mA tDCS
Device: Sham tDCS — One session of sham stimulation.
  Arms: Sham tDCS

SUMMARY:
This is a randomized double-blind sham controlled systematic investigation to understand the importance of the brain region that controls the tongue and the submental muscle region on perceived appetite. The results of this study can have clinical implications for a phenomenon called hyperphagia.

DETAILED DESCRIPTION:
After explaning all the procedure and the scientific aims of the project to participants and completing the informed consent form, each participant will be randomly asked to take part in the experiment while fasting for at least 6 hours or completely sated, to enable an investigation of the role of the basic level of hunger on the effects of brain stimulation on subjective appetite. Different intensities of stimulation (1 mA, 1.5 mA, and sham) will be used in three separate groups, to which participants will be randomly assigned, in a double-blind manner.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight, based on the Body Mass Index (BMI)
* Males and females between 18 and 35

Exclusion Criteria:

* Use of psychoactive drugs
* Presence of metal implants in the brain, skull, scalp or neck
* Use of pacemaker
* Neurological or psychiatric pathologies
* History of severe head injury
* Pregnancy
* Clinical obesity based on BMI

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Change in the subjective rating of appetite | Baseline measurement in the begninning of the experiment before stimulation versus post stimulation, exactly after the stimulation protocol has finished (with an approximate time interval of 1 hour)
  A visual analogue scale (VAS; from 0 meaning not hungry at all, to 100 meaning extremely hungry), will be used to record the perceived level of hunger before and after the stimulation to enable evaluation of the effects of stimulation on perceived appetite.

SECONDARY OUTCOMES:
Change in excitability of the submental muscle region in primary motor cortex | Baseline measurement in the begninning of the experiment before stimulation versus post stimulation, exactly after the stimulation protocol has finished (with an approximate time interval of 1 hour)
  Recording motor evoked potentials from the area of the submental region of the motor cortex in addition to a control site (APB muscle), to allow for comparisons of the amplitude of MEPs before and after stimulation to draw conclusions about the effect of stimulation and its contribution to the potential behavioral modulations of tDCS

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Mario Vicario, PhD, Study Director — University of Messina
Locations (1):
- University of Messina, Messina, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No